CLINICAL TRIAL: NCT04444128
Title: IMPRoving Cardiovascular RiSk Stratification Using T1 Mapping in General populatION
Acronym: IMPReSSION
Status: Recruiting | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Valentina Puentmann, Priv Doz Dr Dr, Johann Wolfgang Goethe University Hospital
Other Study IDs: IMPReSSION Study
Record Dates: First submitted 2020-06-01; First posted 2020-06-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Myocarditis; Heart Failure; Myocardial Fibrosis; Vascular Inflammation; Long COVID Syndrome
Keywords: Inflammation; Remodeling; vascular inflammation
MeSH Terms: conditions — Myocarditis; Heart Failure; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac Imaging — Subjects undergo CMR study with contrast agent (gadobutrol 0.1 mmol/kg; mapping, volumes, function, strain and LGE); transthoracic echocardiography, blood sampling and cardiopulmonary exercise testing.

SUMMARY:
Magnetic properties of myocardial tissue change in the presence of disease. This is detectable in the change of rate of magnetic relaxation, and measurable by T1 and T2 mapping using cardiovascular magnetic resonance (CMR). These markers provide novel quantifiable imaging measures for myocardial tissue characterisation. Despite similar principles, the measurements differ considerably between different sequences, vendors and field strengths, yielding a necessity to establish robust sequence-specific normal ranges, diagnostic accuracy, relationships with clinical characteristics, cardiovascular risk factors, routine cardiac imaging parameters, and prognosis. A further unknown relates to separation between healthy myocardium and subclinical disease in subgroups of patients with suspected cardiac involvement. Examples include patients with possible inflammation, such as in patients with a recent COVID-19 infection or vaccination. Anticipated recruitment of a total of 3000 subjects, with 1500 subjects per field strength (1.5 and 3.0 Tesla).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. 18 years of age and over
3. Absence of a valid clinical indication for CMR, and/or known or clinically relevant cardiac disease

Exclusion Criteria:

* accepted contraindications for a contrast-enhanced CMR study (in line with MRI safety and SmPC for contrast agent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are consecutive asymptomatic healthy subjects or patients from subgroups with known high risk (such as a recent COVID19 infection) with no known or clinically relevant cardiac disease or currently prescribed cardiac medication.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-11-15 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year
  number of deaths
All-cause mortality | 5 years
  number of deaths

SECONDARY OUTCOMES:
Heart Failure Outcome | 1 year and 5 years
  Number of participants with events including death due to heart failure and and hospitalisation due to Heart Failure
Cardiovascular Outcome | 1 year and 5 years
  Number of participants with death due to myocardial infarction, heart failure, arrhythmia or vascular events (pulmonary embolism, aortic dissection, stroke)
Arrhythmia Outcome | 1 year and 5 years
  Number of participants with documented events including sudden cardiac death, appropriate ICD discharge, sustained VT

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Puntmann VO, Carerj ML, Wieters I, Fahim M, Arendt C, Hoffmann J, Shchendrygina A, Escher F, Vasa-Nicotera M, Zeiher AM, Vehreschild M, Nagel E. Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered From Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Nov 1;5(11):1265-1273. doi: 10.1001/jamacardio.2020.3557. PMID 32730619
- [Result] Puntmann VO, Martin S, Shchendrygina A, Hoffmann J, Ka MM, Giokoglu E, Vanchin B, Holm N, Karyou A, Laux GS, Arendt C, De Leuw P, Zacharowski K, Khodamoradi Y, Vehreschild MJGT, Rohde G, Zeiher AM, Vogl TJ, Schwenke C, Nagel E. Long-term cardiac pathology in individuals with mild initial COVID-19 illness. Nat Med. 2022 Oct;28(10):2117-2123. doi: 10.1038/s41591-022-02000-0. Epub 2022 Sep 5. PMID 36064600
- [Result] Shchendrygina A, Ka MM, Rodriguez C, Alsoufi S, Hoffmann J, Kumar P, Carerj ML, Vanchin B, Holm N, Karyou A, Ganbat M, Nagel E, Puntmann VO. Subclinical patterns of cardiac involvement by transthoracic echocardiography in individuals with mild initial COVID-19. Sci Rep. 2025 Jan 30;15(1):3772. doi: 10.1038/s41598-025-85221-w. PMID 39885199
- See also: Related Info — http://www.cardiac-imaging.org/impression-study.html